CLINICAL TRIAL: NCT06642870
Title: Rare Autoimmune Self-management Programme Development
Acronym: RAISE
Status: Recruiting | Type: Observational
Sponsor: University of the West of England (Other)
Collaborators: University of Leeds (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS number 336948
Record Dates: First submitted 2024-09-09; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Systemic Lupus Erthematosus; Systemic Vasculitis; Inflammatory Myositis; Systemic Sclerosis (SSc); ANCA Associated Vasculitis (AAV); Sjogren Syndrome
Keywords: Rare autoimmune rheumatic diseases; Self-management; Psychological support
MeSH Terms: conditions — Systemic Vasculitis; Scleroderma, Systemic; Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Sjogren's Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study involves a series of focus groups followed by a cross-sectional survey of people with RAIRDs: Systemic lupus erythematosus, systemic vasculitis, inflammatory myositis, systemic sclerosis, Sjogren's syndrome, ANCA-associated vasculitis.
  Interventions: Other: Non-interventional study

INTERVENTIONS:
Other: Non-interventional study — The study will consist of focus groups and a large scale patient survey

SUMMARY:
The rare autoimmune rheumatic diseases (RAIRDs) are life-long multi-system diseases that are life or organ threatening. RAIRDs can impair quality of life similar to chronic diseases such as heart failure. The aim of the study is to explore content and structure of a support programme for people with RAIRDs in focus groups and survey meetings.

DETAILED DESCRIPTION:
This project aims to provide self-management and psychological support for people with rare autoimmune rheumatic diseases. The first aim is to ensure that the support provided is relevant for all people, through reaching people who may not have been involved in research before. The second aim is to get agreement for the content and structure of this support from people with these diseases and healthcare teams across the UK.

The rare autoimmune rheumatic diseases include systemic lupus erythematosus, vasculitis, scleroderma, myositis and Sjogren's syndrome. They can affect people of any age and can be fatal. They often have a negative impact on peoples' quality of life (social, work and family life).

Information was gathered from six online meetings with groups of people who have these conditions. People wanted to know the truth about their disease and treatment, alongside help adapting to living with a rare and serious disease. A survey of NHS rheumatology departments shows that the majority (80%) do not provide support to help patients deal with the impact of living with one of these diseases.

Firstly, six groups of patients in total (2 each in Bristol, Weston-Super-Mare and Leeds) will be organised with the help of community groups. Focus groups will help gather a range of views regarding support needs.

Secondly, a UK-wide patient survey of support needs will be conducted, translated into the ten most spoken languages in the UK. Paper versions will be available in NHS rheumatology departments, and an online version will be shared through patient charities.

Lastly, survey results and group responses will be used to build a picture of the type of support needed and how to achieve this in practice. The research team will present the results to the patient partners involved, charities, NHS management and healthcare professionals asking the question: How can support be achieved for patients with rare rheumatic diseases within the current NHS? The research team will then make changes to the support programme based on the feedback received.

The researcher leading the patient and public involvement will work closely with community groups. The three patient partners, who have lived experience (one vasculitis and two lupus patients) will work within the research team throughout the life of the project and will take part in all decision making. A group will be formed from patient participants and patient research partners to help design the next steps of the support programme together.

Patient research partners will help design how the outcome of this research will be shared with healthcare professionals and patients. This will include publications, lay summaries shared by patient organisations and presentations at conferences and community events.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of a rare rheumatic condition made by hospital doctor or secondary care: including lupus, systemic vasculitis, myositis, Sjogren syndrome (participant self-report)
2. Ability to give informed consent (with translation support if needed)

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited via NHS Rheumatology sites, local or national registries, community centres, social media and networks for each focus group in Bristol, Weston and Leeds
Sampling Method: Non-Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Self-management/efficacy PROM | In year 1 during the cross-sectional survey
  This study involves qualitative research. The focus group phase will not include outcome measurements. In the cross-sectional survey participants will be asked two questions about self-management and efficacy descriptively to describe the cohort/people who take part

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Robson, Principal Investigator — University of the West of England
Locations (1):
- University of the West of England/ Bristol Royal Infirmary, Bristol, United Kingdom

IPD SHARING:
Plan to Share IPD: No
This is not an interventional study

REFERENCES:
- [Result] Petrocchi V, Visintini E, De Marchi G, Quartuccio L, Palese A. Patient Experiences of Systemic Lupus Erythematosus: Findings From a Systematic Review, Meta-Summary, and Meta-Synthesis. Arthritis Care Res (Hoboken). 2022 Nov;74(11):1813-1821. doi: 10.1002/acr.24639. Epub 2022 Jul 13. PMID 34133081
- [Result] Fernandez M, Alarcon GS, Calvo-Alen J, Andrade R, McGwin G Jr, Vila LM, Reveille JD; LUMINA Study Group. A multiethnic, multicenter cohort of patients with systemic lupus erythematosus (SLE) as a model for the study of ethnic disparities in SLE. Arthritis Rheum. 2007 May 15;57(4):576-84. doi: 10.1002/art.22672. PMID 17471524
- [Result] Jolly M. How does quality of life of patients with systemic lupus erythematosus compare with that of other common chronic illnesses? J Rheumatol. 2005 Sep;32(9):1706-8. PMID 16142864
- [Result] Bowman SJ, St Pierre Y, Sutcliffe N, Isenberg DA, Goldblatt F, Price E, Hamburger J, Richards A, Rauz S, Regan M, Rigby S, Jones A, Mulherin D, Clarke AE. Estimating indirect costs in primary Sjogren's syndrome. J Rheumatol. 2010 May;37(5):1010-5. doi: 10.3899/jrheum.090734. Epub 2010 Apr 1. PMID 20360188
- [Result] Quaresma M, Coleman MP, Rachet B. 40-year trends in an index of survival for all cancers combined and survival adjusted for age and sex for each cancer in England and Wales, 1971-2011: a population-based study. Lancet. 2015 Mar 28;385(9974):1206-18. doi: 10.1016/S0140-6736(14)61396-9. Epub 2014 Dec 3. PMID 25479696
- [Result] Flossmann O, Berden A, de Groot K, Hagen C, Harper L, Heijl C, Hoglund P, Jayne D, Luqmani R, Mahr A, Mukhtyar C, Pusey C, Rasmussen N, Stegeman C, Walsh M, Westman K; European Vasculitis Study Group. Long-term patient survival in ANCA-associated vasculitis. Ann Rheum Dis. 2011 Mar;70(3):488-94. doi: 10.1136/ard.2010.137778. Epub 2010 Nov 24. PMID 21109517
- [Result] Gaubitz M. Epidemiology of connective tissue disorders. Rheumatology (Oxford). 2006 Oct;45 Suppl 3:iii3-4. doi: 10.1093/rheumatology/kel282. PMID 16987829
- See also: Related Info — https://rairda.org/